CLINICAL TRIAL: NCT01811953
Title: Bioequivalence of Empagliflozin/Metformin Fixed Dose Combination Tablets Compared to Single Tablets Administered Together in Healthy Male and Female Volunteers Under Fed and Fasted Conditions (an Open-label, Randomised, Single-dose, Crossover Study)
Brief Title: Equivalence of Resorption of Empagliflozin/Metformin Administered as Combination Tablet Compared With Empagliflozin/Metformin as Single Tablets Administered Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.8; 2012-005156-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (6):
- 1 Empagliflozin/Metformin (T) (Experimental): fixed-dose-combination tablet, oral with 240 ml water under fasted conditions
  Interventions: Drug: Empagliflozin/Metformin
- 2 Empagliflozin/Metformin (T) (Experimental): fixed-dose-combination tablet, oral with 240 ml water under fed conditions
  Interventions: Drug: Empagliflozin/Metformin
- 3 Empagliflozin + Metformin (R) (Experimental): tablets, oral with 240 ml water under fasted conditions
  Interventions: Drug: Empagliflozin; Drug: Metformin
- 4 Empagliflozin + Metformin (R) (Experimental): tablets, oral with 240 ml water under fed conditions
  Interventions: Drug: Empagliflozin; Drug: Metformin
- 5 Empagliflozin/Metformin (T) (Experimental): fixed-dose-combination tablet, oral with 240 ml water under fed conditions
  Interventions: Drug: Empagliflozin/Metformin
- 6 Empagliflozin + Metformin (R) (Experimental): tablets, oral with 240 ml water under fed conditions
  Interventions: Drug: Empagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Empagliflozin — medium dose oral administration
  Arms: 4 Empagliflozin + Metformin (R)
Drug: Metformin — oral administration
  Arms: 4 Empagliflozin + Metformin (R)
Drug: Empagliflozin — low dose of Empagliflozin oral administration
  Arms: 6 Empagliflozin + Metformin (R)
Drug: Empagliflozin/Metformin — low dose of Empagliflozin
  Arms: 5 Empagliflozin/Metformin (T)
Drug: Metformin — oral administration
  Arms: 6 Empagliflozin + Metformin (R)
Drug: Empagliflozin/Metformin — medium dose of Empagliflozin oral administration
  Arms: 2 Empagliflozin/Metformin (T)
Drug: Empagliflozin — medium dose oral administration
  Arms: 3 Empagliflozin + Metformin (R)
Drug: Metformin — oral administration
  Arms: 3 Empagliflozin + Metformin (R)
Drug: Empagliflozin/Metformin — medium dose of Empagliflozin oral administration
  Arms: 1 Empagliflozin/Metformin (T)

SUMMARY:
Bioequivalence of an empagliflozin/metformin (FDC) tablet compared with single tablets of two strength of empagliflozin and metformin (Part I) under fasted and under fed conditions and bioequivalence of empagliflozin/metformin (FDC) tablet compared with single tablets empagliflozin and metformin under fed conditions (Part II).

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.8.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Emp/Met Fasted / Emp+Met Fasted / Emp/Met Fed / Emp+Met Fed: fixed-dose-combination (FDC) tablet under fasted conditions first; then free dose combination tablets under fasted conditions; then FDC tablet under fed conditions; then free dose combination tablets under fed conditions
  Empagliflozin (Emp): 12.5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
- Emp/Met Fed / Emp+Met Fed / Emp/Met Fasted / Emp+Met Fasted: fixed-dose-combination (FDC) tablet under fed conditions first; then free dose combination tablets under fed conditions; then FDC tablet under fasted conditions; then free dose combination tablets under fasted conditions
  Empagliflozin (Emp): 12.5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
- Emp+Met Fasted / Emp/Met Fasted / Emp+Met Fed / Emp/Met Fed: free dose combination tablets under fasted conditions first; then fixed-dose-combination (FDC) tablet under fasted conditions; then free dose combination tablets under fed conditions; then FDC tablet under fed conditions
  Empagliflozin (Emp): 12.5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
- Emp+Met Fed / Emp/Met Fed / Emp+Met Fasted / Emp/Met Fasted: free dose combination tablets under fed conditions first; then FDC tablet under fed conditions; then free dose combination tablets under fasted conditions; then fixed-dose-combination (FDC) tablet under fasted conditions
  Empagliflozin (Emp): 12.5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
- Low Dose Emp: Emp/Met / Emp+Met: fixed-dose-combination tablet under fed conditions first; then free dose combination tablets under fed conditions
  Empagliflozin (Emp): 5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
- Low Dose Emp: Emp+Met / Emp/Met: free dose combination tablets under fed conditions first; then fixed-dose-combination tablet under fed conditions
  Empagliflozin (Emp): 5 mg; Metformin (Met): 1000 mg (oral with 240 ml water)
Period: Overall Study
Arm/Group | Emp/Met Fasted / Emp+Met Fasted / Emp/Met Fed / Emp+Met Fed | Emp/Met Fed / Emp+Met Fed / Emp/Met Fasted / Emp+Met Fasted | Emp+Met Fasted / Emp/Met Fasted / Emp+Met Fed / Emp/Met Fed | Emp+Met Fed / Emp/Met Fed / Emp+Met Fasted / Emp/Met Fasted | Low Dose Emp: Emp/Met / Emp+Met | Low Dose Emp: Emp+Met / Emp/Met
Started | 6 | 6 | 6 | 6 | 12 | 12
Completed | 6 | 6 | 6 | 5 | 11 | 11
Not Completed | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Emp/Met Fasted / Emp+Met Fasted / Emp/Met Fed / Emp+Met Fed | Emp/Met Fed / Emp+Met Fed / Emp/Met Fasted / Emp+Met Fasted | Emp+Met Fasted / Emp/Met Fasted / Emp+Met Fed / Emp/Met Fed | Emp+Met Fed / Emp/Met Fed / Emp+Met Fasted / Emp/Met Fasted | Low Dose Emp: Emp/Met / Emp+Met | Low Dose Emp: Emp+Met / Emp/Met | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (6.7) | 26.5 (9.7) | 28.5 (9.5) | 33.2 (7.1) | 32.8 (9.8) | 32.3 (9.6) | 31.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 4 | 7 | 7 | 25
  Male | 3 | 3 | 5 | 2 | 5 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity, Empagliflozin
Description: AUC0-inf: area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for Empagliflozin
Time Frame: 1 hour (h) before first drug administration and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30 min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: Pharmacokinetic set (PKS): included all subjects of the TS who provided at least one observation for at least one primary PK endpoint and who did not have a protocol violation relevant to the evaluation of Pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 22 | 23
nmol*h/L | 2810 (19.3) | 2580 (20.4) | 2760 (20.0) | 2570 (20.7) | 988 (16.2) | 927 (18.0)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratio of the geometric means (gMean), test/reference, for the primary endpoints using an acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; Geometric mean ratio = 102.55, 90% CI 2-sided [99.531 to 105.653], Standard Error of Mean 1.017 — The geometric mean ratio was calculated as the geometric mean of '1 Empagliflozin/Metformin (T)' divided by the geometric mean of '3 Empagliflozin + Metformin (R)'
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 98.88, 90% CI 2-sided [94.879 to 103.059], Standard Error of Mean 1.024 — The geometric mean ratio was calculated as the geometric mean of '2 Empagliflozin/Metformin (T)' divided by the geometric mean of '4 Empagliflozin + Metformin (R)'
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 106.00, 90% CI 2-sided [102.728 to 109.386], Standard Error of Mean 1.018 — The geometric mean ratio was calculated as the geometric mean of '5 Empagliflozin/Metformin (T)' divided by the geometric mean of '6 Empagliflozin + Metformin (R)'

2. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity, Metformin
Description: AUC0-inf: area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for Metformin
Time Frame: as for outcome 1
Population: PKS: included all subjects of the TS who provided at least one observation for at least one primary PK endpoint and who did not have a protocol violation relevant to the evaluation of Pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 21 | 23
ng*h/mL | 10400 (23.0) | 9220 (26.4) | 11000 (26.8) | 9140 (22.9) | 9080 (32.7) | 9060 (26.7)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 96.13, 90% CI 2-sided [91.25 to 101.26], Standard Error of Mean 1.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 99.34, 90% CI 2-sided [92.56 to 106.62], Standard Error of Mean 1.04 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean difference = 100.81, 90% CI 2-sided [95.74 to 106.14], Standard Error of Mean 1.03 — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point, Empagliflozin
Description: AUC0-tz: area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point for Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 22 | 23
nmol*h/L | 2770 (19.2) | 2530 (20.1) | 2720 (20.0) | 2510 (20.2) | 962 (16.3) | 903 (18.2)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 102.33, 90% CI 2-sided [99.315 to 105.430], Standard Error of Mean 1.017 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 98.82, 90% CI 2-sided [94.784 to 103.037], Standard Error of Mean 1.024 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 105.98, 90% CI 2-sided [102.730 to 109.329], Standard Error of Mean 1.018 — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma, Empagliflozin
Description: Cmax: maximum measured concentration of the analyte in plasma for Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 22 | 23
nmol/L | 379 (23.7) | 276 (24.8) | 375 (27.3) | 258 (28.5) | 108 (16.9) | 103 (14.5)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 102.12, 90% CI 2-sided [96.255 to 108.351], Standard Error of Mean 1.035 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0082, ANOVA; Geometric mean ratio = 106.52, 90% CI 2-sided [95.863 to 118.353], Standard Error of Mean 1.063 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 104.352, 90% CI 2-sided [99.152 to 110.224], Standard Error of Mean 1.031 — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma, Metformin
Description: Cmax: maximum measured concentration of the analyte in plasma for Metformin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 21 | 23
ng/mL | 1580 (26.9) | 1160 (17.8) | 1680 (25.8) | 1180 (21.2) | 1180 (23.8) | 1150 (24.8)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANOVA; Geometric mean ratio = 94.87, 90% CI 2-sided [88.931 to 101.210], Standard Error of Mean 1.038 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 97.97, 90% CI 2-sided [92.339 to 103.935], Standard Error of Mean 1.035 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 102.95, 90% CI 2-sided [97.166 to 109.082], Standard Error of Mean 1.034 — [estimate comment as in outcome 1, analysis 3]

6. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point, Metformin
Description: AUC0-tz: area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point for Metformin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Number analyzed (Participants) | 23 | 24 | 24 | 22 | 21 | 23
ng*h/mL | 10100 (21.3) | 8960 (24.5) | 10700 (24.1) | 8930 (22.5) | 8870 (30.8) | 8850 (26.3)
Statistical Analysis 1: Comparison: 1 Empagliflozin/Metformin (T) vs 3 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 94.89, 90% CI 2-sided [89.80 to 100.26], Standard Error of Mean 1.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2 Empagliflozin/Metformin (T) vs 4 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 99.31, 90% CI 2-sided [92.14 to 107.03], Standard Error of Mean 1.04 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 5 Empagliflozin/Metformin (T) vs 6 Empagliflozin + Metformin (R); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; Geometric mean ratio = 100.74, 90% CI 2-sided [95.77 to 105.96], Standard Error of Mean 1.03 — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: From first trial medication intake until next intake or the end-of-trial visit, 10 days
Description: Adverse Evens were reported for all patients who received the specific treatment.
Arm/Group | 1 Empagliflozin/Metformin (T) | 2 Empagliflozin/Metformin (T) | 3 Empagliflozin + Metformin (R) | 4 Empagliflozin + Metformin (R) | 5 Empagliflozin/Metformin (T) | 6 Empagliflozin + Metformin (R)
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 6/23 | 6/24 | 4/24 | 6/24 | 9/23 | 10/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Empagliflozin/Metformin (T) (N=23) | 2 Empagliflozin/Metformin (T) (N=24) | 3 Empagliflozin + Metformin (R) (N=24) | 4 Empagliflozin + Metformin (R) (N=24) | 5 Empagliflozin/Metformin (T) (N=23) | 6 Empagliflozin + Metformin (R) (N=23)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 2 | 1 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 4 | 4 | 6
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No